CLINICAL TRIAL: NCT06687941
Title: A Multi-center, Open-label, Dose Escalation and Expansion, Phase 1 Study to Evaluate the Tolerability, Safety and Pharmacokinetics of AST-201 in Patients With GPC3-positive Advanced Solid Tumors
Brief Title: A Study to Evaluate the Tolerability, Safety, and PK of AST-201 in Patients With GPC3-positive Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aptamer Sciences, Inc. (Industry)
Collaborators: CHA University (Other); National Cancer Center, Korea (Other Government); Samsung Medical Center (Other); Severance Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AST-201-01
Record Dates: First submitted 2024-11-05; First posted 2024-11-14 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Neoplasms; Carcinoma, Hepatocellular; Carcinoma, Non-Small-Cell Lung; Liver Neoplasms
Keywords: Glypican-3 (GPC3); GPC3-positive advanced solid tumors; AST-201; Aptamer-drug conjugate; Hepatocellular carcinoma (HCC); Advanced solid tumors; Metastatic; Dose Escalation and Expansion
MeSH Terms: conditions — Neoplasms; Carcinoma, Hepatocellular; Carcinoma, Non-Small-Cell Lung; Liver Neoplasms; Simpson-Golabi-Behmel syndrome; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AST-201 (Experimental)
  Interventions: Drug: AST-201

INTERVENTIONS:
Drug: AST-201 — AST-201 is administered intravenously on Days 1, 8, and 15 of each 28-day cycle, followed by a one-week rest period. Dosing is repeated until DLT or disease progression is occurred.

SUMMARY:
This is the first in human trial clinical study of AST-201 in patients with GPC3-positive advanced solid tumors. This study aims to evaluate the safety, tolerability, pharmacokinetic properties, and preliminary efficacy of AST-201 across various tumor types.

DETAILED DESCRIPTION:
AST-201 is a novel aptamer drug conjugate (ApDC) investigational agent with demonstrated preclinical efficacy in GPC3-positive tumor models. This Phase 1 clinical study aims to investigate the safety, tolerability, and preliminary efficacy of AST-201, targeting GPC3-positive advanced solid tumors. The study consists of two parts: Phase 1a and Phase 1b.

In Phase 1a, AST-201 will be administered in a dose escalating manner across cohorts of patients to determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D). In this dose-escalation phase, patients will receive AST-201 as a single agent, with safety, tolerability, and pharmacokinetic (PK) profiles assessed. In Phase 1b, patients will receive AST-201 at the RP2D across specific GPC3-positive tumor types to further explore safety and efficacy. This expansion phase focuses on assessing anti-tumor efficacy and overall safety in a broader patient population. Data collected from this study will support future clinical development of AST-201 in GPC3-positive advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria

* Male and female aged ≥19 years
* Histologically and/or cytologically diagnosed as the advanced recurrent solid tumor
* GPC3-positive confirmed by IHC test
* At least 1 measurable or non-measurable but evaluable lesion as defined per RECIST v1.1 (modified RECIST for hepatocellular carcinoma)
* ECOG performance status of 0 or 1
* Life expectancy at least 12 weeks
* Adequate hematologic, hepatic, renal, and heart/coagulation function
* Child-Pugh Class of A for HCC

Exclusion Criteria

* Subjects with ischemic heart disease
* Subjects with anti-tumor treatment within 4 weeks
* Subjects with comorbidities such as uncontrolled hypertension, heart failure, etc.
* Pregnant or potentially pregnant and lactating woman

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | 4 weeks

SECONDARY OUTCOMES:
Pharmacokinetics (PK) | Cycle 1, Days 1-2 (cycle is 28 days)
  Maximum Plasma Concentration (Cmax)
Pharmacokinetics (PK) | Cycle 1, Days 1-2 (cycle is 28 days)
  Time to Reach Maximum Plasma Concentration (Tmax)
Pharmacokinetics (PK) | Cycle 1, Days 1-2 (cycle is 28 days)
  Area Under the Curve (AUC)
Pharmacokinetics (PK) | Cycle 1, Days 1-2 (cycle is 28 days)
  Clearance Rate
Pharmacokinetics (PK) | Cycle 1, Days 1-2 (cycle is 28 days)
  Half-Life (t1/2)
Preliminary Antitumor Efficacy | Baseline through the end of each 28-day cycle, up to 6 months.
  Objective Response Rate (ORR) is defined as the proportion of subjects with the best overall response (BOR) assessed as complete response (CR) and partial response (PR). ORR assessed by the Investigator and evaluated according to RECIST 1.1 criteria.
Preliminary Antitumor Efficacy | Baseline through the end of each 28-day cycle, up to 6 months.
  Disease Control Rate (DCR) is defined as the proportion of subjects with the BOR assessed as CR, PR, or stable disease (SD). DCR assessed by the Investigator and evaluated according to RECIST 1.1 criteria.
Preliminary Antitumor Efficacy | Baseline through the end of each 28-day cycle, up to 6 months.
  Duration of Response (DOR) is defined as the period from the initial assessment date confirming CR or PR to disease progression (PD) or death. DOR assessed by the Investigator and evaluated according to RECIST 1.1 criteria.
Preliminary Antitumor Efficacy | Baseline through the end of each 28-day cycle, up to 6 months.
  Time to Progression (TTP) is defined as the period from the initial administration of the investigational product (IP) to disease progression (PD). TTP assessed by the Investigator and evaluated according to RECIST 1.1 criteria.
Preliminary Antitumor Efficacy | Baseline through the end of each 28-day cycle, up to 6 months.
  Progression-Free Survival (PFS) is defined as the period from the initial administration of the IP to disease progression (PD) or death. PFS assessed by the Investigator and evaluated according to RECIST 1.1 criteria.
Preliminary Antitumor Efficacy | Baseline through the end of each 28-day cycle, up to 6 months.
  Overall Survival(OS) is defined as the period from the initial administration of the IP to death.

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - National Cancer Center, Korea, Gyeonggi-do
  - CHA Bundang Medical Center, Seongnam
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No